CLINICAL TRIAL: NCT03783299
Title: Assessing the Effectiveness of Targeted Active Case Detection Among High Risk Populations in Southern Lao PDR
Brief Title: Targeted Active Case Detection Among High Risk Populations in Southern Lao Peoples Democratic Republic
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Center for Malariology, Parasitology, and Entomology (Unknown); The National Institute of Public Health (Unknown); Health Poverty Action (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: 17-22577; A124497 (Other Grant/Funding Number: Bill & Melinda Gates Foundation)
Record Dates: First submitted 2018-11-30; First posted 2018-12-21 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Plasmodium Falciparum Malaria
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artemether, Lumefantrine Drug Combination; Primaquine

STUDY DESIGN:
Intervention Model Description: The study is employing a split-plot community-randomized controlled trial design, with peer navigator test and treat randomized at the health center catchment level, and village-based test and treat randomized at the village level within health center catchment areas (HCCA).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Village-based MTAT (Experimental): Intervention: For all households in intervention villages, after obtaining informed consent, MTAT will be conducted with all household members aged 18 months and older.
  The MTAT team will test each individual using both a standard RDT and HS-RDTs. Positive cases will be treated with age-appropriate doses of Artemether-lumefantrine (AL) and Primaquine Phosphate (SLD-PQ)
  Interventions: Diagnostic Test: Standard RDT and HS-RDT; Drug: Artemether-lumefantrine; Drug: Primaquine Phosphate
- Peer navigator-led FTAT (Experimental): Intervention: Peer navigators will actively seek non-village based HRPs in forested areas, rice fields and plantations, and any other non-permanent settlements within target health center catchment areas, and conduct FTAT among all consenting individuals.
  The Peer Navigators will test each individual using both a standard RDT and HS-RDT. Positive cases will be treated with age-appropriate doses of Artemether-lumefantrine (AL) and Primaquine Phosphate (SLD-PQ)
  Interventions: Diagnostic Test: Standard RDT and HS-RDT; Drug: Artemether-lumefantrine; Drug: Primaquine Phosphate

INTERVENTIONS:
Diagnostic Test: Standard RDT and HS-RDT — All household members (residents and temporary visitors) aged 18 months and older will be invited to participate in an RDT and blood collection component. After consenting, the MTAT team will capture axillary temperature, and test each individual using both a standard RDT (SD Bioline Pf/Pv RDT) and HS-RDT (SD Bioline Malaria Ag P.f High Sensitive Cat# 05FK140)
  Other Names: SD Bioline Alere Malaria Ag Pf High Sensitive Cat #05FK140; SD Bioline Pf/Pv RDT
  Arms: Village-based MTAT
Diagnostic Test: Standard RDT and HS-RDT — All individuals will be invited to participate in an RDT and blood collection component. Informed consent will be obtained from all participants. After consenting, the PNs will capture axillary temperature, and test each individual using both a standard RDT (SD Bioline Pf/Pv RDT) and HS-RDT (SD Bioline Alere Malaria Ag Pf High Sensitive Cat #05FK140). Dried blood spots (DBS) will also be collected on all HRPs if deemed feasible.
  Other Names: SD Bioline Alere Malaria Ag Pf High Sensitive Cat #05FK140; SD Bioline Pf/Pv RDT
  Arms: Peer navigator-led FTAT
Drug: Artemether-lumefantrine — If found positive by standard RDT or HS-RDT, treatment will be administered, and women of reproductive age will be assessed as outlined in the protocol. All individuals who have provided informed consent, test positive by either HS-RDT or standard RDT, are ≥18 months old, are not pregnant or breastfeeding, and who do not have symptoms associated with severe malaria or another severe illness, will be offered an age-appropriate course of AL (age-specific blister packages) and SLD-PQ according to national treatment guidelines.
  Other Names: Coartem
Drug: Primaquine Phosphate — If found positive by standard RDT or HS-RDT, treatment will be administered, and women of reproductive age will be assessed as outlined in the protocol. All individuals who have provided informed consent, test positive by either HS-RDT or standard RDT, are ≥18 months old, are not pregnant or breastfeeding, and who do not have symptoms associated with severe malaria or another severe illness, will be offered an age-appropriate course of AL (age-specific blister packages) and SLD-PQ according to national treatment guidelines.
  Other Names: Primaquine

SUMMARY:
This study assesses the effectiveness of targeted active case detection among high-risk populations in Southern Lao Peoples Democratic Republic (PDR). The investigators hypothesize that active case detection using the next generation of HRP-2 rapid diagnostic tests (RDTs) can help bridge gaps in identification of high-risk asymptomatic individuals with low density parasitemia, allowing for targeting of this reservoir and thereby reducing transmission. The investigators hypothesize that active case detection (testing and treating positive cases) with these RDTs will lead to a reduction in P. falciparum transmission.

DETAILED DESCRIPTION:
This study is the second phase of work in Champasak Province, Southern Lao PDR, building off a formative phase of work that characterized the demographics, occupations, migratory patterns, health-seeking behaviors, and social networks of mobile and migrant populations (MMPs) in four target districts. This phase of the study now aims to determine the effectiveness, cost-effectiveness, acceptability, and feasibility of proactive targeted test-and-treat activities using high-sensitivity malaria rapid diagnostic tests (HS-RDTs) for reducing Plasmodium falciparum malaria transmission in Champasak Province among (1) village residents and (2) mobile and migrant populations (MMPs) and other high-risk populations (HRPs).

The study will specifically assess the role of HS-RDTs, a diagnostic test that offers potentially ~10-fold greater sensitivity than standard RDTs, in active case detection at both the village-level and in forest-going HRPs for decreasing prevalence and incidence of P. falciparum in target areas. The effectiveness of these interventions will be compared independently and in combination against areas with no study interventions (standard of care) over the course of implementation (planned for October 2017 - November 2018).

The two main study interventions are mass test and treat (MTAT) using HS-RDTs in village-based populations, and peer navigator (PN) led focal test and treat (FTAT) using HS-RDTs in forest based HRPs. Primary outcomes will include PCR-based P. falciparum prevalence at endline. Following a baseline cross-sectional survey in November-December 2017, the interventions will consist of 3 rounds of MTAT spaced throughout the year, with potential to reduce to 2 based upon initial prevalence estimates, and ongoing FTAT by PNs among forest and forest-fringe HRPs, with the primary evaluation to be conducted through an end-line cross-sectional survey in November 2018.

ELIGIBILITY:
Village Based MTAT

Inclusion Criteria

* All household members 18 months of age and older.
* Study participants include those in the 14 selected health center catchment areas within the four target districts in Champasak Province, Southern Lao PDR; Moulapamook, Panthampone, Sanamsaboun, and Soukhuma.
* Members of households who have provided informed consent will be included for blood samples collection and treatment for identified malaria cases if meeting the appropriate criteria.

Exclusion Criteria

* Household members less than 18 months of age will be excluded.
* Any individuals under the age of 18 months will be excluded from RDT testing and blood collection.

Peer Naviagtor-Led FTAT

Inclusion Criteria

* All persons 15 years and older who have spent at least one night outside a formal village in the past one month.
* Individuals must be 18 years and older and willing and able to provide consent to be included in the peer navigator or study staff focus group discussions and key informant interviews
* Study participants include those in the 14 selected health center catchment areas within the four target districts in Champasak Province, Southern Lao PDR; Moulapamook, Panthampone, Sanamsaboun, and Soukhuma
* High-risk populations in forested areas, rice field regions, plantations and any informal settlements
* Individuals travelling into the HCCA who are willing and sufficiently able to communicate with PNs to assess their eligibility

Exclusion criteria

- Individuals under the age of 18 will be excluded from peer navigator or study staff focus group discussions and key informant interviews.

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39968 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Community-level PCR-based P. falciparum prevalence in sampled villages | 4 months
  This is defined as the proportion of individuals >18 months old with P. falciparum infection (detected by PCR) out of all individuals >18 months tested within the 2017 and 2018 surveys.The effectiveness of the interventions will be assessed as P. falciparum prevalence via PCR at end-line (post only) using generalized linear mixed effects models with separate random intercepts to allow for clustering within villages and health center catchments. The binomial distribution will be used to analyze prevalence outcomes (logistic regression)
HS-RDT-based test positivity rate in village-based and forest-based samples | 6 months
  This is defined as the proportion of all individuals tested by HS-RDT at each round of the MTAT interventions or during routine FTAT, with a positive HS-RDT, among the population older than 18 months.The HS-RDT and RDT test positivity rates will be estimated for the MTAT villages during each intervention round. This will be done as soon as data on RDT and HS-RDT results are available, which would be expected to be one month following each round. Differences in prevalence measures at each round will be assessed using a χ2 test, as well as logistic regression models to account for potential confounding factors.
Village-based population coverage of test and treat interventions | 3 months
  This indicator will be measured in two ways for each round of village MTAT. Operational program coverage is defined as the proportion of individuals ≥18 months old and households visited and offered the MTAT interventions within the target areas. Effective program coverage is defined as the proportion of individuals (≥18 months old) that agreed to participate in the MTAT intervention among all individuals ≥18 months old eligible to participate in the intervention in the target population
Community-level confirmed P. falciparum malaria parasite incidence | 1 year
  This is defined as the number of total and confirmed outpatient (OPD) malaria confirmed and suspected cases per person per year for each village, as ascertained from the health facility registers, utilizing village population size estimates for the exposure denominator. Data pertaining to this outcome will be analyzed on an intention-to-treat basis. Monthly counts of confirmed malaria cases from the health facility registers will be linked to villages and analyzed in a time series Poisson or negative binomial model with random intercepts at the health center catchment and village levels.

SECONDARY OUTCOMES:
Serology | 2 months
  Seropositivity to a panel of standard malaria parasite antigens for P. falciparum and P. vivax (including merozoite surface protein-1 (MSP-1) and apical membrane antigen-1 (AMA-1), will be used to examine both recent and medium-term exposures. These data will also be mapped used captured global positioning system (GPS) coordinates to examine serological hotspots. Finally, novel antigens will also be used to further explore any differences in parasite exposure between study arms. Vector exposure may also be explored using antigens to anopheline salivary proteins.
Cost and cost effectiveness | 12 months
  For the costing portion of the study, the cost per case investigation conducted, cost per additional positive case identified using FTAT in village- and forest-based HRPs, and the cost per case actively detected per person screened during screen and treat. The cost-effectiveness of screen and treat will also be compared between village-based activities and peer-navigator led testing.
Sensitivity and specificity of HS-RDTs | 6 months
  The P. falciparum prevalence from all individuals tested with HS-RDTs will be compared with parallel results from standard RDTs (all field testing activities) and to subsequent PCR-based testing (cross-sectional survey, FTAT and MTAT subset). In the latter case, the PCR-based result will serve as the gold standard for all comparisons. Sensitivity and specificity and receiver operating curve (ROC) analyses will be conducted to assess the performance of the HS-RDTs in field situations, and in the presence of mixed-species infections. DBS will be collected for cross-sectional survey, FTAT and MTAT.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Bennett, MA, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Centre for Marialogy, Parasitology, and Entomology, Vientiane, Laos

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with any parties outside of the study team.

REFERENCES:
- [Background] Tiono AB, Ouedraogo A, Ogutu B, Diarra A, Coulibaly S, Gansane A, Sirima SB, O'Neil G, Mukhopadhyay A, Hamed K. A controlled, parallel, cluster-randomized trial of community-wide screening and treatment of asymptomatic carriers of Plasmodium falciparum in Burkina Faso. Malar J. 2013 Feb 27;12:79. doi: 10.1186/1475-2875-12-79. PMID 23442748
- [Background] Mosha JF, Sturrock HJ, Greenhouse B, Greenwood B, Sutherland CJ, Gadalla N, Atwal S, Drakeley C, Kibiki G, Bousema T, Chandramohan D, Gosling R. Epidemiology of subpatent Plasmodium falciparum infection: implications for detection of hotspots with imperfect diagnostics. Malar J. 2013 Jul 1;12:221. doi: 10.1186/1475-2875-12-221. PMID 23815811
- [Background] Cook J, Xu W, Msellem M, Vonk M, Bergstrom B, Gosling R, Al-Mafazy AW, McElroy P, Molteni F, Abass AK, Garimo I, Ramsan M, Ali A, Martensson A, Bjorkman A. Mass screening and treatment on the basis of results of a Plasmodium falciparum-specific rapid diagnostic test did not reduce malaria incidence in Zanzibar. J Infect Dis. 2015 May 1;211(9):1476-83. doi: 10.1093/infdis/jiu655. Epub 2014 Nov 26. PMID 25429102
- [Background] Hustedt J, Canavati SE, Rang C, Ashton RA, Khim N, Berne L, Kim S, Sovannaroth S, Ly P, Menard D, Cox J, Meek S, Roca-Feltrer A. Reactive case-detection of malaria in Pailin Province, Western Cambodia: lessons from a year-long evaluation in a pre-elimination setting. Malar J. 2016 Mar 1;15:132. doi: 10.1186/s12936-016-1191-z. PMID 26931488
- [Background] Parker DM, Landier J, von Seidlein L, Dondorp A, White L, Hanboonkunupakarn B, Maude RJ, Nosten FH. Limitations of malaria reactive case detection in an area of low and unstable transmission on the Myanmar-Thailand border. Malar J. 2016 Nov 25;15(1):571. doi: 10.1186/s12936-016-1631-9. PMID 27887652
- [Background] Hoyer S, Nguon S, Kim S, Habib N, Khim N, Sum S, Christophel EM, Bjorge S, Thomson A, Kheng S, Chea N, Yok S, Top S, Ros S, Sophal U, Thompson MM, Mellor S, Ariey F, Witkowski B, Yeang C, Yeung S, Duong S, Newman RD, Menard D. Focused Screening and Treatment (FSAT): a PCR-based strategy to detect malaria parasite carriers and contain drug resistant P. falciparum, Pailin, Cambodia. PLoS One. 2012;7(10):e45797. doi: 10.1371/journal.pone.0045797. Epub 2012 Oct 1. PMID 23049687
- [Background] Cotter C, Sturrock HJ, Hsiang MS, Liu J, Phillips AA, Hwang J, Gueye CS, Fullman N, Gosling RD, Feachem RG. The changing epidemiology of malaria elimination: new strategies for new challenges. Lancet. 2013 Sep 7;382(9895):900-11. doi: 10.1016/S0140-6736(13)60310-4. Epub 2013 Apr 15. PMID 23594387
- [Background] World Health Organization. Strategy for malaria elimination in the Greater Mekong Subregion: 2015-2030 [Internet]. Geneva: Global Malaria Program, WHO; 2015. Available: http://iris.wpro.who.int/bitstream/handle/10665.1/10945/9789290617181_eng.pdf
- [Background] World Health Organization Regional Office for South-East Asia (SEARO). Approaches for mobile and migrant populations in the context of malaria multi-drug resistance and malaria elimination in the Greater Mekong Subregion [Internet]. Thailand; 2016. Available: http://apps.who.int/iris/bitstream/10665/204351/2/Approaches_%20mobile_migrant_populations.pdf
- [Background] Center for Malariology, Parasitology, and Entomology, Lao PDR. Lao PDR Malaria National Strategic Plan 2016-2020. Vientiane, Lao PDR: Ministry of Health, Lao PDR; 2015.
- [Derived] Lover AA, Dantzer E, Hocini S, Estera R, Rerolle F, Smith JL, Hwang J, Gosling R, Yukich J, Greenhouse B, Jacobson J, Phetsouvanh R, Hongvanthong B, Bennett A. Study protocol for a cluster-randomized split-plot design trial to assess the effectiveness of targeted active malaria case detection among high-risk populations in Southern Lao PDR (the AcME-Lao study). Gates Open Res. 2019 Dec 17;3:1730. doi: 10.12688/gatesopenres.13088.1. eCollection 2019. PMID 32118199

DOCUMENTS (1):
  • Study Protocol (2017-11-05): https://cdn.clinicaltrials.gov/large-docs/99/NCT03783299/Prot_000.pdf